CLINICAL TRIAL: NCT05618717
Title: Surpoint Algorithm for Improved Guidance of Ablation for Ventricular Tachycardia in Patients With Ischemic and Non-Ischemic Cardiomyopathy
Brief Title: Surpoint Algorithm for Improved Guidance of Ablation for Ventricular Tachycardia
Acronym: SURFIRE-VT
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Henry Huang, Primary Investigator, Rush University Medical Center
Other Study IDs: 21011101
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Surpoint Index Guided Ablation Group: Maximum Radiofrequency delivery duration cannot exceed Surpoint Index of 550
  Interventions: Device: Radiofrequency Ablation
- Conventional Ablation Group: Operator determined ablation duration regardless of Surpoint Index Value
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — Radiofrequency Ablation using irrigated ablation catheter

SUMMARY:
Vistag SurPoint is a proprietary module that generates a numerical tag index which can be used as multiparametric lesion quality marker to guide ablation in the clinical setting for ablation of atrial arrhythmias. SurPoint tag index has studied to guide ablation of ventricular arrhythmias, such as premature ventricular complexes, but its effectiveness and safety for ablation of Ventricular Tachycardia in patient with Ischemic and Non-Ischemic Cardiomyopathies is not well established.

In this single center prospective observation registry, a ventricular ablation strategy utilizing radiofrequency delivery duration cut off determined by a maximum Surpoint index value of 550 will be compared to conventional operator determined duration of radiofrequency delivery based on combination of time (i.e. 30, 60, 90, and 120 seconds), magnitude of impedance drop, attenuation of abnormal electrograms, and achieving non-capture with high-output pacing after ablation.

The Surpoint Tag Index Ablation group will be matched with a control group of patients undergoing VT ablation using the conventional time-based radiofrequency strategy and the patients in this group will be selected using propensity matching based on relevant baseline patient and clinical characteristic variables.

Primary outcomes of interest: Recurrence of sustained ventricular tachycardia or Internal Cardiac Defibrillator Therapy.

Secondary outcomes of interest: Hospitalization for ventricular tachycardia, repeat ablation procedures, all-cause mortality, acute procedural complications, rate of steam pops during ablation procedures

Follow up: Up to 24 months after ablation procedure. Follow up will be obtained by office visits and device interrogation reports.

ELIGIBILITY:
Inclusion Criteria:

* Structural Heart Disease: Ischemic or Non-Ischemic Cardiomyopathy
* Sustained Monomorphic Ventricular Tachycardia documented by ECG or CIED interrogation

Exclusion Criteria:

* If clinical ventricular arrhythmia is predominantly PVCs, polymorphic ventricular tachycardia, or ventricular fibrillation
* Myocardial infarction or Cardiac Surgery within 6 months
* Severe mitral regurgitation
* Stroke or TIA within 6 months
* Prior Ventricular Tachycardia Ablation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: History of Ischemic or non-ischemic cardiomyopathy with sustained ventricular tachycardia
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence Event of Sustained Ventricular Tachycardia or ICD therapy | 2 years
  Composite outcome of sustained ventricular tachycardia (episode lasting > 30 seconds detected by ICD) or ventricular tachycardia episode treated successfully by ICD therapy (Including ventricular tachycardia episodes terminated by ATP or ICD shock in < 30 seconds based programmed detection/treatment ICD settings)

SECONDARY OUTCOMES:
Hospitalization for Ventricular Tachycardia | 2 yearr
  Outcome of hospitalization for primary admission diagnosis of ventricular tachycardia with or without ICD treatment
All-Cause Mortality | 2 years
  Outcome of death after ablation procedure from cardiovascular or non-cardiovascular cause
Redo Ventricular Tachycardia Ablation Procedure | 2 years
  Outcome of repeat ablation procedure for sustained ventricular tachycardia or appropriate ICD therapy after index ventricular tachycardia ablation procedure
Procedural Complications | 7 days
  Outcome of rate of complications with 7 days of ventricular tachycardia ablation procedure including but not limited to bleeding, death, pericardial effusion, cardiac tamponade, stroke, arterial thromboemblism, steam pops, thrombus formation, cardiogenic shock, phrenic nerve paralysis, congestive heart failure)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Huang, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Casella M, Gasperetti A, Gianni C, Zucchelli G, Notarstefano P, Al-Ahmad A, Burkhardt JD, Soldati E, Della Rocca D, Catto V, Majocchi B, Carbucicchio C, Bongiorni MG, Dello Russo A, Natale A, Tondo C. Ablation Index as a predictor of long-term efficacy in premature ventricular complex ablation: A regional target value analysis. Heart Rhythm. 2019 Jun;16(6):888-895. doi: 10.1016/j.hrthm.2019.01.005. Epub 2019 Jan 4. PMID 30616020
- [Background] Gasperetti A, Sicuso R, Dello Russo A, Zucchelli G, Saguner AM, Notarstefano P, Soldati E, Bongiorni MG, Della Rocca DG, Mohanty S, Carbucicchio C, Duru F, Di Biase L, Natale A, Tondo C, Casella M. Prospective use of ablation index for the ablation of right ventricle outflow tract premature ventricular contractions: a proof of concept study. Europace. 2021 Jan 27;23(1):91-98. doi: 10.1093/europace/euaa228. PMID 33063099
- [Background] Sciacca V, Vogler J, Eitel C, Kuck KH, Tilz RR, Heeger CH. Ablation index-guided catheter ablation of incessant ventricular tachycardia originating from the anterolateral papillary muscle. Clin Res Cardiol. 2022 May;111(5):588-591. doi: 10.1007/s00392-021-01923-x. Epub 2021 Nov 1. No abstract available. PMID 34724088
- [Background] Larsen T, Du-Fay-de-Lavallaz JM, Winterfield JR, Ravi V, Rhodes P, Wasserlauf J, Trohman RG, Sharma PS, Huang HD. Comparison of ablation index versus time-guided radiofrequency energy dosing using normal and half-normal saline irrigation in a porcine left ventricular model. J Cardiovasc Electrophysiol. 2022 Apr;33(4):698-712. doi: 10.1111/jce.15379. Epub 2022 Jan 30. PMID 35048448